CLINICAL TRIAL: NCT07166679
Title: Effect of Apical Third Enlargement to Different Taper and Master Apical Preparation Size on Periapical Healing and Postoperative Pain After Primary Single Sitting Non Surgical Root Canal Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sahil
Record Dates: First submitted 2025-08-25; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Asymptomatic Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP A HAVING MASTER APICAL FILE SIZE # 25 (Experimental): group a is further dived into 3 further subgroup a1 2% taper a2 4% taper a3 6% taper
  Interventions: Procedure: root canal treatment with 2% taper; Procedure: root canal treatment with 4% taper; Procedure: root canal treatment with 6 %taper
- GROUP B HAVING MASTER APICAL FILE SIZE # 30 (Experimental): GROUP B is further divide into 3 further subgroup b1 2% taper b2 4 % taper b3 6 % taper
  Interventions: Procedure: root canal treatment with 2% taper; Procedure: root canal treatment with 4% taper; Procedure: root canal treatment with 6 %taper
- GROUP C HAVING MASTER APICAL FILE SIZE # 35 (Experimental): GROUP C is further divide into 3 subgroups c1 2 % taper c2 4 % taper c3 6 % taper
  Interventions: Procedure: root canal treatment with 2% taper; Procedure: root canal treatment with 4% taper; Procedure: root canal treatment with 6 %taper

INTERVENTIONS:
Procedure: root canal treatment with 2% taper — root canal treatment with 2%taper
Procedure: root canal treatment with 4% taper — root canal treatment with 4 %taper
Procedure: root canal treatment with 6 %taper — root canal treatment with 6 %taper

SUMMARY:
To Determine Effect Of Apical Third enlargement To Different Taper And Master Apical Preparation Size On Periapical Healing And Postoperative Pain After Primary Single Sitting Non Surgical Root Canal Treatment : A Randomized Clinical Trial

DETAILED DESCRIPTION:
The primary goal of endodontic therapy is to eradicate microbial infection within the root canal system and prevent reinfection. Thorough debridement and disinfection of the apical third are crucial, as this region serves as a reservoir for residual microorganisms.

Till date, only four clinical trials have analysed the effect of apical canal preparation size on treatment outcomes. Out of the four clinical trials one retrospective in nature, Hoskinson study no improvement in radiographic and clinical outcome with an increase in the master apical file .

Souza (2012) conducted clinical trial in necrotic pulp and concluded that apical third enlargement does not alter endodontic treatment outcomes.

Saini (2012) stated that enlarging the canal three sizes beyond the first apical binding file is sufficient.

Fatima (2021) found that preparing the apical region in two sizes larger the initial apical binding file (IABF) with a 4% taper is inadequate, leading to significantly lower success rates compared to larger preparation sizes and greater tapers .

In both studies( Fatima and saini ) determination of apical enlargement size was based on the IABF (initial apical binding file). There was no mention of master apical size in different groups. Also the taper of apical one third was different in both these studies.Both master apical size and preparation taper can influence root canal shaping in apical third Various in-vitro studies suggest that increasing the taper has no significant effect on bacterial reduction.

According to Plotino(2014) the difference in the taper of the instruments did not result in different levels of disinfection in the apical region. They observed that amount of infected residual dentin & the smear layer in the apical third of root canals were not significantly affected by preparations with 0.04 or 0.06 tapers when the apical diameter remained the same. Other studies examining bacterial reduction and different tapers agree with these results (Alimadadi, 2021; Usta 2023).

There is no impact on bacteria reduction when using different tapers with the same apical size #25 in the preparation of the mesial root canals of mandibular molars. ( Macedo, 2024) while clinical study by Fatima suggests that increasing the taper promotes better periapical healing. In Fatima study, a significantly high success rate was observed with apical preparation 2 sizes larger than the IABF and a 6% taper compared with the same preparation size with a 4%taper (92.8% vs 57.1%.).Till date there is no clinical study that combined the effect of different master apical file size and different taper on outcome of primary nonsurgical root canal treatment. Therefore, the present study was designed as a randomized clinical trial to examine the effect of apical third enlargement to different taper and master apical preparation size on periapical healing and postoperative pain after primary single sitting non surgical root canal treatment

Primary objective :

To evaluate and compare the radiographic outcome of periapical healing after primary non surgical single sitting root canal with different tapers and different master apical file size

Secondary objective :

To assess the post operative pain using VAS scale, postoperatively every 24 hours for 1 week after primary nonsurgical single sitting root canal treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age of either sex
2. Asymptomatic teeth having pulpal necrosis with apical periodontitis in a mandibular molar (no response to EPT or cold test)
3. Radiographic evidence of periapical radiolucency corresponding to a periapical index (PAI) score >/=3 in mesial root of mandibular molars

Exclusion Criteria:

1. Patients who were medically compromised
2. Patients with initial apical binding file (IABF) size more than 20
3. Pregnancy; lactation & contraceptives.
4. Positive history of antibiotic use within the past month or required antibiotic premedication for dental treatment (including infective endocarditis or pros thetic joint prophylaxis -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2027-04-18 (Estimated)

PRIMARY OUTCOMES:
periapical healing using the Periapical index score | 12 month follow up
  Description: Periodical status will be assessed in periapical radiograph • Periapical status will be checked according to periapical index given by Orstavik
  * Scoring of periapical radiolucency of each tooth will be done according to the following 5 point scale (PAI score)
  * Score 1- Normal periapical structure
  * Score 2- Small changes in bone structure
  * Score 3- Changes in bone structure with some mineral loss
  * Score 4- Periodontitis with well-defined radiolucent area
  * Score 5- Severe periodontitis with exacerbating features
  Time Frame: 12MONTHS

SECONDARY OUTCOMES:
post operative pain | Baseline and at 24 hours, Day 2, Day 3, Day 4, Day 5, Day 6 and Day 7 after the treatment
  Post Operative Pain To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score100 means maximum pain. To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score 100 means maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Dr shweta MITTAL, MDS, Principal Investigator — PDIDS ROHTAK
Locations (1):
- Pgids Rohtak, Rohtak, India

IPD SHARING:
Plan to Share IPD: No